CLINICAL TRIAL: NCT05478304
Title: Left Atrial Appendage Exclusion for Prophylactic Stroke Reduction Trial
Acronym: LeAAPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CP-2021-05
Record Dates: First submitted 2022-07-15; First posted 2022-07-28 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2024-10

CONDITIONS: Ischemic Stroke; Systemic Embolism
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment (Experimental): LAAE using the AtriClip concomitant to and at the time of planned cardiac surgery
  Interventions: Device: AtriClip LAA Exclusion System
- Control (No Intervention): No LAAE concomitant to and at the time of planned cardiac surgery

INTERVENTIONS:
Device: AtriClip LAA Exclusion System — LAAE using the AtriClip concomitant to and at the time of planned cardiac surgery
  Arms: Treatment

SUMMARY:
This trial is a prospective, randomized, multicenter, multinational, blinded, superiority trial. The objective of this trial is to evaluate the effectiveness of left atrial appendage exclusion (LAAE) for the prevention of ischemic stroke or systemic arterial embolism in subjects undergoing cardiac surgery who have risk factors for atrial fibrillation and ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age
* Documentation of any of the following clinical criteria:

  * CHA2DS2-VASc ≥ 4 with age ≥ 65
  * CHA2DS2-VASc ≥ 4 with significant left atrium enlargement or elevated NT-proBNP
  * CHA2DS2-VASc = 3 with age ≥ 75
  * CHA2DS2-VASc = 3 with significant left atrium enlargement or elevated NT-proBNP
  * CHA2DS2-VASc score = 2 with age ≥ 65 and significant left atrium enlargement or elevated NT-proBNP

Exclusion Criteria:

* Clinically significant atrial fibrillation or atrial flutter:

  * Anytime in the past and
  * Documented by an electrocardiographic recording and
  * Episode lasting 6 minutes or longer1*
* Prior procedure involving opening the pericardium or entering the pericardial space
* Prior LAA occlusion, exclusion, or removal (surgical or percutaneous)
* Planned cardiac surgical procedure using non-sternotomy approaches

  o Partial sternotomies will be allowed.
* Patients whose planned procedure is a heart transplant or implantation of any ventricular assist devices
* Active endocarditis
* Active systemic infection at the time of cardiac surgery requiring antibiotics, including known SARS-CoV2 infections regardless of symptoms
* Known allergy to Nitinol or nickel sensitivity
* Known medical condition with expected survival of less than 1 year
* Other comorbidities that in the investigator's opinion make the subject unsuitable candidate to complete the protocol required visits.
* Current enrollment in an investigation or trial or an investigational devices or investigational drug that would interfere with this trial.
* Mental impairment or other psychiatric conditions which may not allow the patient to understand the nature, significance, and scope of the trial.
* Pregnancy
* Known severe symptomatic carotid disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6573 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | Common termination point (median follow-up for 5 years)
  Time to the first occurrence of ischemic stroke or systemic arterial embolism as adjudicated by the Clinical Events Committee (CEC), or any procedure wherein the LAA was excluded, occluded, or amputated following the index procedure.
Primary Safety Endpoint | 30 days post index procedure
  Occurrence of at least one of the following events assessed through 30 days post index procedure:
  * Pericardial effusion requiring percutaneous or surgical treatment
  * Major bleeding attributable to index surgical procedure
  * Deep sternal wound infection
  * Myocardial infarction

SECONDARY OUTCOMES:
Powered Secondary Effectiveness endpoint | Common termination point (median follow-up for 5 years)
  Time to the first occurrence of ischemic stroke or systemic arterial embolism

CONTACTS AND LOCATIONS:
Overall Officials: Richard Whitlock, MD, Study Chair — McMaster University
Locations (143):
- United States (107):
  - Heart Center Research / Huntsville Hospital, Huntsville, Alabama
  - HonorHealth Shea Scottsdale Healthcare, Scottsdale, Arizona
  - St. Bernard's Heart & Vascular, Jonesboro, Arkansas
  - CHI St. Vincent, Little Rock, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Memorial Care Long Beach Medical Center, Long Beach, California
  - Keck Medical Center of USC, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Sutter Sacramento Hospital, Sacramento, California
  - Stanford University, Stanford, California
  - University of Colorado, Boulder, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - HCA Florida JFK Hospital, Atlantis, Florida
  - HealthPark Medical Center, Fort Myers, Florida
  - University of Florida Hospital, Gainesville, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Baptist Health Jacksonville, Jacksonville, Florida
  - Baptist Health South Florida, Miami, Florida
  - Advent South, Orlando, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tampa General Hospital, Tampa, Florida
  - Baycare Health System, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Wellstar - Kennestone, Marietta, Georgia
  - St. Luke's Regional Medical Center, Boise, Idaho
  - Portneuf Medical Center, Idaho Falls, Idaho
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Memorial Hospital (SIU Medicine), Springfield, Illinois
  - Ascension St. Vincent, Carmel, Indiana
  - Franciscan, Indianapolis, Indiana
  - Mercy Medical Center, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - St. Luke's Hospital, Kansas City, Kansas
  - Kansas University Medical Center, Kansas City, Kansas
  - Baptist Health, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Norton Healthcare, Louisville, Kentucky
  - University of Louisville Health / Jewish Hospital, Louisville, Kentucky
  - Novant Presbyterian Hospital, Louisville, Kentucky
  - Our Lady of the Lake Hospital, Baton Rouge, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Corewell Health East, Royal Oak, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Trinity Health (formerly St. Joesph Mercy), Ypsilanti, Michigan
  - Mercy Medical Center, Coon Rapids, Minnesota
  - Abbott Northwestern / Minneapolis Heart, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Midwest Heart and Vascular (HCA), Kansas City, Missouri
  - St. Lukes Hospital, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Nebraska Methodist, Omaha, Nebraska
  - The Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Robert Woods Johnson Medical School, New Brunswick, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - North Shore University Hospital (Northwell), Manhasset, New York
  - St. Francis Hospital, Roslyn, New York
  - St. Joseph Hospital, Syracuse, New York
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - WakeMed Health & Hospitals, Raleigh, North Carolina
  - Wake Forest Baptist, Winston-Salem, North Carolina
  - TriHealth / Bethesda North Hospital, Cincinnati, Ohio
  - Christ Hospital / Lindner Research Center, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State Medical Center, Columbus, Ohio
  - Riverside Methodist, Columbus, Ohio
  - The Toledo Hospital (Promedica), Toledo, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - UPMC Pinnacle, Harrisburg, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Health System, Pittsburgh, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Jackson Madison County General, Jackson, Tennessee
  - Centennial Medical Center (TriStar), Nashville, Tennessee
  - Ascension St. Thomas West, Nashville, Tennessee
  - UT Dell Medical School, Austin, Texas
  - HCA Medical City Dallas, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Baylor Heart Hospital - Plano, Plano, Texas
  - Trinity Mother Frances (CHRISTUS), Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - Inova Fairfax Medical, Falls Church, Virginia
  - Sentara Hospitals & Sentara Medical Group, Norfolk, Virginia
  - Swedish Heart and Vascular Research, Seattle, Washington
  - Charleston Area Medical Center (CAMC), Charleston, West Virginia
  - West Virginia University, Morgantown, West Virginia
  - Columbia St. Mary's, Milwaukee, Wisconsin
  - Aspirus Hospital, Wausau, Wisconsin
- Australia (3):
  - Gold Coast University Hospital, Southport, Queensland
  - Victorian Heart Hospital and Monash University, Clayton, Victoria
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
- Austria (2):
  - Medical University Hospital Graz, Graz, Styria
  - Medical University Vienna, Vienna
- Belgium (2):
  - University Hospitals UZ Leuven, Leuven, Brabant
  - UZ Brussels, Jette, Brussels Capital
- Canada (14):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - New Brunswick Heart Centre, Saint John, New Brunswick
  - Queen Elizabeth II - Nova Scotia Health, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - IUCPQ Hosptial Laval, Québec
- CKTCH Brno, Brno, Czechia
- Germany (6):
  - University Heart Venter Freiburg Bad Krozingen, Freiburg im Breisgau, Baden-Wurttemberg
  - Rhön-Klinikum Campus Bad Neustadt, Bad Neustadt an der Saale, Bavaria
  - Deutsches Herzzentrum der Charité, Berlin, Brandenburg
  - Bad Rothefelde Schüchtermann-Klinik, Bad Rothenfelde, Lower Saxony
  - University Heart and Vascular Center Hamburg, Hamburg
  - Albertinen Krankenhaus, Hamburg
- Waikato Hospital-Hamilton, Hamilton, Waikato Region, New Zealand
- Spain (2):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Clinico San Carlos, Madrid
- United Kingdom (5):
  - Northern General Hospital, Sheffield, Great Britain
  - St. Bartholomew's Hospital, London, Greater London
  - The James Cook University Hospital, Middlesbrough, North Yorkshire
  - The Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands
  - Royal Papworth Hospital, Cambridge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whitlock RP, McCarthy PM, Gerdisch MW, Ramlawi B, Alexander JH, Sultan I, Rose DZ, Healey JS, Sharma YA, Belley-Cote EP, Connolly SJ. The left atrial appendage exclusion for prophylactic stroke reduction (LEAAPS) trial: Rationale and design. Am Heart J. 2025 Jun;284:94-102. doi: 10.1016/j.ahj.2024.10.006. Epub 2024 Oct 11. PMID 39395566